CLINICAL TRIAL: NCT01795924
Title: An Open-Label, Phase 1/2 Study of PD-616 and Low-dose Cytarabine in Patients With Untreated or Relapsed/Refractory Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Safety and Efficacy Study of PD-616 Plus Cytarabine to Treat Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Acronym: AML/MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty of patient enrollment
Sponsor: Biosuccess Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT12-US-AML-a
Record Dates: First submitted 2013-02-13; First posted 2013-02-21 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD-616 plus low-dose Cytarabine (Experimental): Patients will receive low-dose cytarabine (20 mg/m2) subcutaneously (SC) once daily (QD), followed by a 1-hour intravenous (IV) infusion of PD-616 for 5 consecutive days during Week 1 (D1 to D5) and Week 2 (D8 to D12) of a 28-day treatment cycle. Cytarabine is to be administered approximately 30 minutes before PD-616. In Phase 1 part, the starting dose of PD-616 is 0.0875 mg/m2, with sequential increments of 0.0375 mg/m2, to 0.125, and 0.1625 mg/m2. The dose of PD-616 to be administered in Phase 2 part will be the maximum tolerated dose (MTD)determined from Phase 1 part of the study.
  Interventions: Drug: PD-616

INTERVENTIONS:
Drug: PD-616 — Patients may continue treatment through 1 year post-C1D1 or until withdrawal of consent or development of any toxicity meeting the definition of Dose-Limiting Toxicity or progressive disease, whichever occurs first.
  Other Names: TPA; 12-O-Tetra-Decanoyl-Phorbol-13-Acetate

SUMMARY:
The purpose of this study is to determine whether PD-616 in combination with low-dose Cytarabine is safe and effective in the treatment of untreated or relapsed/refractory acute myelogenous leukemia (AML) or high-risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Protocol RT12-US-AML-a is a 2-part, Phase 1/2, multi-center, open-label, dose-escalation study of PD-616 in combination with low-dose cytarabine in patients with AML or high-risk MDS not eligible for standard therapy.

Part 1 of this study (Phase 1 portion) employs a sequential group-dose escalation design to determine the DLT and MTD of PD-616 in combination with low-dose cytarabine (primary objective). The safety and PK profiles as well as the preliminary efficacy of PD-616 in combination with cytarabine also will be examined (secondary objectives). Approximately 21 patients are planned to be enrolled in Part 1.

After provision of written informed consent, patients are to be evaluated for study eligibility during the Screening period which should be within 14 days before the first day of study drug administration (Cycle 1, Day 1 [C1D1]; Baseline). Patients who are determined to be eligible, based on Screening assessments, will be enrolled in the study on C1D1, which is the first day of study drug administration.

Part 2 of this study (Phase 2 portion) will commence with approval of the Safety Review Committee (SRC) after identification of the MTD, or if the MTD is not established, the maximum feasible dose has been evaluated in Part 1. Twelve additional patients will be enrolled and treated with PD-616 at the MTD (or other biologically relevant dose) in combination with low-dose cytarabine according to the same schedule as in Part 1. The safety profile, PK, and efficacy of the study drug combination will be further investigated in Part 2 of this study.

Each cycle of treatment consists of a treatment period (D1 through D12) and a rest period (D13 through D28). During the treatment period, patients are required to return to the study center on D1 through D5 and D8 through D12 for study drug to be administered and evaluations to be performed. During the rest period, patients are required to return to the study center at least once a week for study evaluations. In addition, patients are required to be evaluated for peripheral blasts by flow cytometry in the last week of each cycle (D22 to D28) and to receive bone marrow examination in the last week (D22 to D28) of C1. Patients with evidence of complete response (CR) in peripheral blood by flow cytometry are to have a repeat bone marrow examination performed to confirm CR.

All patients are to attend the Study Drug Discontinuation Visit within 3 days after discontinuing study drug. Thereafter, patients will enter the post-study period and be followed monthly (±3 days), starting 30±3 days after last study drug administration, through 1 year post-C1D1. During the post-study period, patients who discontinue for reasons other than progressive disease (PD) also will have follow-up blood samples collected for evaluation of changes in the percentage of blasts every month until PD or receipt of alternative therapy, whichever occurs first, up to 1 year post-C1D1. During the post-study period, patients with evidence of CR in peripheral blood by flow cytometry are to have a repeat bone marrow examination performed to confirm CR.

ELIGIBILITY:
Inclusion Criteria:

* Patient has newly diagnosed AML and refuses or is not eligible for treatment with aggressive chemotherapy and/or SCT; OR AML and has relapsed or been refractory to prior therapy; OR High-risk MDS, defined as IPSS intermediate-2 (INT-2) or IPSS high-risk, and refuses or is not eligible for standard or aggressive chemotherapy and SCT or prior experimental therapies; OR High-risk MDS, defined as IPSS INT-2 or IPSS high risk, and has failed or been refractory to deoxyribonucleic acid (DNA) hypomethylating agents (azacitidine or decitabine), lenalidomide, standard/aggressive chemotherapy, SCT, or prior experimental therapies.
* Has a bone marrow examination performed within 14 days before baseline (C1D1).
* Has an ECOG performance status score of 0 to 2.
* Aged between 18 and 75 years, inclusive.
* Has a life expectancy of ≥3 months.
* Has the following laboratory parameters within 7 days before baseline (C1D1):Serum creatinine ≤2 mg/dL; Total bilirubin ≤2.0 mg/dL; Alanine transaminase (ALT) or aspartate transaminase (AST) <3.0×the upper limit of normal (ULN); Left ventricular ejection fraction (LVEF) >40%; Forced expiratory volume in 1 second (FEV1) >60% of predicted.
* If a female of child-bearing potential, has a negative serum pregnancy test result within 14 days before baseline and agrees to abstain from heterosexual intercourse or use a barrier method for contraception from 14 days before baseline (C1D1) through 30 days after the last study drug dose.
* If male, agrees to use a latex condom during any sexual contact with a female of child-bearing potential.
* Able to understand and willing to provide written informed consent.

Exclusion Criteria:

* Has received prior treatment with PD-616 or low-dose cytarabine.
* Has received chemotherapy (except hydroxyurea), biological therapy, radiotherapy or investigational therapy within 4 weeks before baseline (C1D1).
* Has active central nervous system (CNS) involvement (documented by radiologic lesions and/or malignant cells in the cerebrospinal fluid [CSF]).
* Has acute promyelocytic leukemia (APL, FAB M3).
* Has another active systemic malignancy treated with chemotherapy within 12 months before baseline (C1D1).
* Has known human immunodeficiency virus (HIV) infection.
* Has active graft-versus-host disease (GVHD).
* Has uncontrolled active infection of any kind. (Patients with infections controlled by active antibiotic treatment are eligible).
* Has significant renal or hepatic disease, uncontrolled or severe cardiovascular or pulmonary diseases, or other uncontrolled medical condition that, based on the Investigator's assessment, would compromise the patient's ability to tolerate study treatment or the assessment of treatment response.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The number of dose-limiting toxicities in each cohort of PD-616 in combination of low-dose Cytarabine to determine the maximum tolerated dose of PD-616. | Average 28 days after the first dose of treatment
  Primary outcome measure for the Phase 1 part of the study.
The percentage of patients achieving complete or partial remission after the treatment of PD-616 at the maximum tolerated dose in combination with low-dose Cytarabine. | One year from the first dose of treatment
  Primary outcome measure for Phase 2 part of the study.

SECONDARY OUTCOMES:
The pharmacokinetic profile of PD-616 consisting AUC. | 1 hour before and 20, 40 and 60 minutes during and 0.5, 1, 2, 4, 6, 10 hours after treatment on Day 1 and Day 5 and before treatment on Day 2, Day 3 and Day 4
The pharmacokinetic profile of PD-616 consisting Cmax. | 1 hour before and 20, 40 and 60 minutes during and 0.5, 1, 2, 4, 6, 10 hours after treatment on Day 1 and Day 5 and before treatment on Day 2, Day 3 and Day 4
The pharmacokinetic profile of PD-616 consisting Tmax. | 1 hour before and 20, 40 and 60 minutes during and 0.5, 1, 2, 4, 6, 10 hours after treatment on Day 1 and Day 5 and before treatment on Day 2, Day 3 and Day 4
The pharmacokinetic profile of PD-616 consisting Cmin. | 1 hour before and 20, 40 and 60 minutes during and 0.5, 1, 2, 4, 6, 10 hours after treatment on Day 1 and Day 5 and before treatment on Day 2, Day 3 and Day 4
The proportion of patients experiencing adverse events. | One year from the first dose of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S Stein, MD, Principal Investigator — City of Hope Medical Center; Dianna S. Howard, M.D., Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - University of Kentucky Medical Center, Lexington, Kentucky